CLINICAL TRIAL: NCT00287430
Title: Growth Hormone Use in Adolescents and Adults With Cystic Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: D Hardin not at institution, IRB has no record, no other investigators for study information
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Dana S Hardin (Unknown)
Responsible Party: Principal Investigator, Nancy Rollins, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0102-035
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Growth Hormone; Absorptiometry, Photon

INTERVENTIONS:
Drug: Growth Hormone
Procedure: Whole body Protein Turnover Study
Procedure: Dual Energy X-ray Absorptiometry (DEXA)

SUMMARY:
We hypothesize that the anabolic effects of growth hormone (GH) will improve the clinical status of patients with CF by improving lean body mass, osteopenia, muscle strength, pulmonary function, and quality of life.

We will recruit 40 malnourished CF patients for this 12-month study. All 40 patients will be treated with recombinant human growth hormone (rhGH). Each patient will serve as his/her own control by obtaining medical records for 6 months to 1 year prior to study enrollment or by completing 6 months of study without GH prior to being treated for 1 yr. with GH.

DETAILED DESCRIPTION:
Patients will be treated with growth hormone in the form of Nutropin (a powder formulation that is reconstituted by the patient) or Nutropin AQ (a ready-to-use liquid) for 1 year. Both of these products are manufactured by Genentech, Inc. The starting dose will be 0.006 mg/kg given as a daily subcutaneous (SC) injection. The GH dose will be titrated 1-3 months after GH initiation to maintain blood levels of IGF-1 within the normal range for age and sex. The dose will be increased to a maximum of 0.025 mg/kg daily in adult patients <35 years and to a maximum of 0.0125 mg/kg daily in adult patients > 35 years. Pre-pubertal and adolescent patients will be dosed at 0.3 mg/kg/wk to 0.6 mg/kg/wk.

PROCEDURES:

1. To determine the effect of GH on body weight and lean body mass in CF, weight will be measured at baseline and every three months utilizing the same scale. LBM will be measured at baseline and every six months by dual emission x-ray absorptiometry (DEXA) scan.
2. To determine the effect of GH on protein breakdown and protein synthesis in CF, protein turnover studies will be performed at baseline and every 6 months utilizing the stable isotope C-leucine and mass spectrophotometric analysis.

   Each subject will undergo 30-minute measurements of substrate oxidation and resting energy expenditure using hood indirect calorimetry. Substrate calculations yielding information on glucose oxidation and lipid oxidation will be determined using the methods of de Weir, and results will be correlated with measurements calculated from stable isotope infusion.
3. To determine the effect of GH on hepatic glucose production (HGP) the following study will be performed at baseline and every 6 months.
4. To quantify the portion of hepatic glucose production (HGP) derived from gluconeogenesis and glycogenolysis in the post-absorptive state. We will measure gluconeogenesis using the stable isotope 2H2O and measurement of the incorporation of 2H into the 6th and 2nd carbon of glucose, according to the method of Landau 11.
5. To determine if GH improves the nutritional status of CF patients the following nutritional status indicators will be measured at 6 month intervals: retinal binding protein, transferrin, thyroxine binding prealbumin, albumin, and lipid profile. Additionally, caloric intake and food group consumption will be analyzed by a skilled dietitian from 3-day food journals recorded every six months.
6. To determine if GH improves the clinical condition of CF patients, participants will perform pulmonary function tests, including measurement of PI and PE for estimation of respiratory muscle strength. Additionally, each subject's clinical status will be evaluated at baseline and every 3 months utilizing a modified NIH clinical status scoring system.
7. To determine if GH improves the quality of life of CF patients, participants will complete a 15-minute questionnaire to assess quality of life. This questionnaire entitled "The Cystic Fibrosis Questionnaire" has been recently developed and tested for quality. It is specific for CF patients and has been approved by the National CF Foundation.
8. All patients will have random blood glucose testing per CF Foundation guidelines. If a patient has previously undiagnosed cystic fibrosis related diabetes (CFRD) with or without fasting hyperglycemia (FH), he/she will be treated with insulin for a minimum for 3 months prior to study enrollment. Patients in all other glucose tolerance categories will be allowed to participate in the study Also, patients previously treated with insulin will be allowed to participate if HgbA1C is < 8.5%. If not, the PI will adjust insulin and maximize glycemic control for 3 months before study entry. Any patient who develops CFRD with or without FH will be continued in the study only if he/she will agree to insulin therapy. If a patient refuses insulin therapy, he/she will be discontinued from the study. Patients will continue to be screened for glucose intolerance by measuring random blood glucose and HgbA1C.
9. To further study the sustained effect of GH, all study subjects will be given the option of continuing on GH for an additional year. The same assessments above will be performed every six months for the additional year.

Statistics:

This is a pilot study of 40 subjects. Data will be assessed as mean and standard deviation. Data will then be used to compute a power analysis for a future larger study. Non-treatment data will be compared to treatment data with emphasis on the 12 and 18-month time points. Data from patients who develop CFRD while on the study, if there are any, will be analyzed separately from those who do not develop CFRD.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 40 years
* less than 100% of ideal body weight.

Exclusion Criteria:

* Colonization with Burkholderia cepacia
* pregnancy.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
1) body weight
2) lean body mass.

SECONDARY OUTCOMES:
1) whole body protein turnover
2) hepatic glucose production
3) bone mineral density
4) pulmonary function status
5) quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas